CLINICAL TRIAL: NCT03057639
Title: Adolescent and Young Adult (AYA) Cancers Clinical Model: An Evaluation of the AYA Clinical Care Model by Assessment of Clinical, Psychosocial, and Health Economic Factors Related to AYA Patient Outcomes
Brief Title: Clinical Model in Evaluating Clinical, Psychosocial, and Health Economic Factors in Adolescent and Young Adult Patients With Cancer
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-16-6; NCI-2017-00210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-16-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaires): Patients complete questionnaires at referral, week 4-8, week 10-12, and at the completion of systemic therapy.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies the Adolescent and Young Adult (AYA) Cancers Clinical Model in evaluating clinical, psychosocial, and health economic factors in adolescent and young adult patients with cancer. Studying the Adolescent and Young Adult Cancers Clinical Model may help doctors learn more about the effect of the AYA services on patient care, including clinical (nurse navigation), psychosocial (social work), and economic (financial) areas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide economic understanding of the AYA at University of Southern California (USC) model of care. (Norris)

II. To evaluate the existing AYA at USC program to determine the direct and indirect impact on cost of care. (Norris)

III. To utilize the results of objective (i) to identify cost effectiveness and efficiencies to patient and institution. (Norris)

IV. To identify specific processes within our model of care that can be improved. (Norris)

V. To improve healthcare access to AYA-specific cancer care for patients ages 15-39 served by the Los Angeles County (LAC)+USC oncology pilot clinics. (LAC+USC)

VI. To improve the psychosocial outcome of AYA-specific cancer care patients. (LAC+USC)

VII. To provide AYA specific elements of care routinely and proactively to AYA cancer patients. (LAC+USC)

VIII. To improve care quality through patient satisfaction. (LAC+USC)

IX. To improve resource utilization and care coordination through improved patient navigation through efficiency and patient navigation. (LAC+USC)

OUTLINE:

Patients complete questionnaires at referral, week 4-8, week 10-12, and at the completion of systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer
* ADDITIONAL GRANT SPECIFIC INCLUSION CRITERIA - UNIHEALTH (NORRIS):
* Patients who were diagnosed at USC Norris Comprehensive Cancer Center and Hospital
* Patients who are currently receiving treatment for a primary or secondary tumor at USC Norris Comprehensive Cancer Center and Hospital
* ADDITIONAL GRANT SPECIFIC INCLUSION CRITERIA - QUEENSCARE (LAC + USC):
* Patients who are being seen in sarcoma, gynecologic oncology, or genitourinary clinic at LAC + USC (clinics A2C or 4P1)
* Patients who are currently receiving treatment for a primary or secondary tumor at LAC + USC and who receive oncology care from one of the clinics above
* Patients who are at or below the poverty level

Exclusion Criteria:

* Inability to sign informed assent and/or consent
* Patients who are not receiving chemotherapy and/or radiation therapy for a primary or secondary tumor
* Primary oncology treatment team believes that participation in AYA at USC would not benefit their patient
* ADDITIONAL GRANT SPECIFIC EXCLUSION CRITERIA - UNIHEALTH (NORRIS):
* Patients who are not receiving treatment for a primary or secondary tumor at USC Norris Comprehensive Cancer Center and Hospital
* ADDITIONAL GRANT SPECIFIC EXCLUSION CRITERIA - QUEENSCARE (LAC+USC):
* Patients who are not receiving oncology care for a primary or secondary tumor in sarcoma, gynecologic oncology, or genitourinary clinic at LAC + USC (clinics A2C or 4P1)
* Patients who are above the poverty level

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent and Young Adult (AYA) with cancer who are being seen at the USC/Norris Cancer Center and at LAC+USC Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Clinical care model impact on patient access to AYA specific supportive care as assessed by questionnaires (Norris) | Up to 2 years
  Questionnaire scores will be expressed as median values with 95% confidence intervals.
Clinical care model impact on patient's/health care professional's satisfaction with the AYA at USC program as assessed by questionnaires (LAC+USC) | Up to 2 years
  Questionnaire scores will be expressed as median values with 95% confidence intervals.
Cost of care (Norris) | Up to 2 years
  Direct health care costs analyses will be performed from the Total Costs of Care payer perspective. Direct cost will be estimated from paid claims in the extracted electronic medical records, which will include costs for all health care utilization such as outpatient, procedures, laboratory, emergency room visits, hospitalization, and pharmacy. As the healthcare utilization and costs will likely be extremely skewed, healthcare utilization and cost measures will be estimated by using an econometric model (e.g., a negative binomial regression model for utilization count data [number of services
Incremental cost (Norris) | Up to 2 years
  The incremental cost between AYA enrolled and non-enrolled will be calculated. In addition to estimation the magnitude of the variability attributed to the different sources of variation, we will also generate an influence diagram (also known as tornado diagram) to display which variables exert the most influence on cost driver.
Processes that can be improved (Norris) | Up to 2 years
  Will utilize the prospective data to estimate key aspects of the AYA at USC service. Any variances in the services over time will be utilized to improve quality and reliability care delivery.

SECONDARY OUTCOMES:
Care coordination as assessed by the mean number of supportive care referrals, telephone or email encounters for additional information, educational materials, and or additional interventions provided by the nurse navigator and/or social worker (LAC+USC) | Up to 2 years
  Will be measured using an implementation guide.
Patient continuity of care as assessed by the mean number of visits per patient with the assigned clinic lead physician (LAC+USC) | Up to 2 years
  Will be measured using an implementation guide.
Resource allocation as assessed by the mean number of supportive care referrals and per patient follow-up conducted by the nurse navigator and/or social worker (LAC+USC) | Up to 2 years
  Will be measured using an implementation guide.
Satisfaction of health care staff as assessed by questionnaires (LAC+USC) | Up to 2 years
  Questionnaire scores will be expressed as median values with 95% confidence intervals.
Satisfaction of services as assessed by questionnaires (LAC+USC) | Up to 2 years
  Questionnaire scores will be expressed as median values with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: James Hu, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States